CLINICAL TRIAL: NCT07180277
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Methylprednisolone Sodium Succinate Injection in Patients With Moderate to Severe Traumatic Brain Injury
Brief Title: Methylprednisolone for Moderate to Severe Traumatic Brain Injury
Acronym: ESM-TBI Trail
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhangjiagang First People's Hospital (Other)
Responsible Party: Principal Investigator, Rong Gao, Professor, Zhangjiagang First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZJGSY2025001
Record Dates: First submitted 2025-09-09; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-07

CONDITIONS: Traumatic Brain Injury
Keywords: Methylprednisolone; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- methylprednisolone (Experimental)
  Interventions: Drug: Methylprednisolone (MP)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 2 mg/kg diluted in 100 mL of normal saline (maximum dose 160 mg) , IV once daily for 5 days
  Arms: Placebo
Drug: Methylprednisolone (MP) — 2 mg/kg diluted in 100 mL of normal saline (maximum dose 160 mg) , IV once daily for 5 days
  Arms: methylprednisolone

SUMMARY:
The goal of this clinical trial is to learn if standard-dose methylprednisolone sodium succinate can improve neurological recovery and safety in adults with moderate to severe traumatic brain injury (TBI). The main questions it aims to answer are:

1. Does adding a 5-day course of methylprednisolone improve overall long-term neurological outcome compared with placebo?
2. Does methylprednisolone reduce 6-month mortality or increase the proportion of patients with good neurological recovery?
3. What medical problems do participants experience when receiving methylprednisolone? Researchers will compare methylprednisolone sodium succinate (2 mg/kg/day intravenously for 5 days) with a matching placebo to see if the steroid improves outcomes beyond standard TBI care.

Participants will:

1. Receive either methylprednisolone or placebo once daily for 5 days, added to guideline-directed standard care.
2. Undergo CT scans and neuro-examinations during hospitalization.
3. Return for follow-up visits at 1 month and 6 months after injury for neurological assessments, safety checks, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Patients with moderate-to-severe traumatic brain injury whose Glasgow Coma Scale (GCS) score at admission is 4-12.
* Study drug must be initiated within 12 hours after injury.
* Imaging (CT) demonstrates cerebral contusion, or cerebral contusion with intracerebral hematoma.
* Written informed consent obtained from the subject or legally authorised representative.

Exclusion Criteria:

* Known hypersensitivity to corticosteroids or any contraindication to their use.
* History of diabetes mellitus, or capillary blood glucose <2.8 mmol/L or >22.2 mmol/L.
* Shock at admission (systolic blood pressure <90 mmHg for more than 30 minutes).
* Pregnant or lactating women.
* Participation in another clinical trial within the past 3 months.
* Any condition that, in the investigator's opinion, renders the patient unsuitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of Glasgow Outcome Scale-Extended (GOS-E) scores at 180 days. | 180 days

SECONDARY OUTCOMES:
All-cause mortality | 180 days
Proportion of patients with good neurological outcome (GOS-E 6-8) | 180 days
Incidence of adverse events after treatment | 30 days

REFERENCES:
- [Background] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000
- [Background] Roberts I, Yates D, Sandercock P, Farrell B, Wasserberg J, Lomas G, Cottingham R, Svoboda P, Brayley N, Mazairac G, Laloe V, Munoz-Sanchez A, Arango M, Hartzenberg B, Khamis H, Yutthakasemsunt S, Komolafe E, Olldashi F, Yadav Y, Murillo-Cabezas F, Shakur H, Edwards P; CRASH trial collaborators. Effect of intravenous corticosteroids on death within 14 days in 10008 adults with clinically significant head injury (MRC CRASH trial): randomised placebo-controlled trial. Lancet. 2004 Oct 9-15;364(9442):1321-8. doi: 10.1016/S0140-6736(04)17188-2. PMID 15474134
- [Background] He C, Wang Y, Gong W, Zhang S. Targeted Delivery of Acid-Responsive Rutin Nanoparticles Based on Aldehyde Adsorption for the Treatment of Spinal Cord Injury in Rats. ACS Biomater Sci Eng. 2025 Apr 14;11(4):2192-2202. doi: 10.1021/acsbiomaterials.5c00038. Epub 2025 Apr 1. PMID 40167167
- [Background] Chen X, Chai Y, Wang SB, Wang JC, Yue SY, Jiang RC, Zhang JN. Risk factors for corticosteroid insufficiency during the sub-acute phase of acute traumatic brain injury. Neural Regen Res. 2020 Jul;15(7):1259-1265. doi: 10.4103/1673-5374.272611. PMID 31960811
- [Background] Zhang B, Bai M, Xu X, Yang M, Niu F, Gao F, Liu B. Corticosteroid receptor rebalancing alleviates critical illness-related corticosteroid insufficiency after traumatic brain injury by promoting paraventricular nuclear cell survival via Akt/CREB/BDNF signaling. J Neuroinflammation. 2020 Oct 25;17(1):318. doi: 10.1186/s12974-020-02000-2. PMID 33100225
- [Background] Liu Z, Yang Y, He L, Pang M, Luo C, Liu B, Rong L. High-dose methylprednisolone for acute traumatic spinal cord injury: A meta-analysis. Neurology. 2019 Aug 27;93(9):e841-e850. doi: 10.1212/WNL.0000000000007998. Epub 2019 Jul 29. PMID 31358617
- [Background] Zhang Y, Xiao S, Zhu L, Gan X, Huang Y, Dan F, Chen J, Zhou R, Tang W, Liu J, Liu Z. Effect of Low-dose Methylprednisolone in Promoting Neurological Function Recovery After Spinal Cord Injury: Clinical and Animal Studies. Spine (Phila Pa 1976). 2025 Jul 15;50(14):965-974. doi: 10.1097/BRS.0000000000005269. Epub 2025 Jan 29. PMID 39876698
- [Background] Zheng C, Li R, Shen C, Guo F, Fan D, Yang L, Zhang L, Chen A, Chen Y, Chen D, Zi W, Guo C, Nguyen TN, Albers GW, Campbell BCV, Qiu Z, Hu Z. Methylprednisolone as Adjunct to Thrombectomy for Acute Intracranial Internal Carotid Artery Occlusion Stroke: Post Hoc Secondary Analysis of the MARVEL Randomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2459945. doi: 10.1001/jamanetworkopen.2024.59945. PMID 39964685
- [Background] Wang B, Zhang Q, Liu C, Chen X. Counteracting immunodepression by extracellular matrix hydrogel to promote brain tissue remodeling and neurological function recovery after traumatic brain injury. Biomaterials. 2025 Jul;318:123181. doi: 10.1016/j.biomaterials.2025.123181. Epub 2025 Feb 8. PMID 39970603